CLINICAL TRIAL: NCT06761768
Title: Efficacy of Combining Corticosteroid Injections and Extracorporeal Shockwave Therapy in Patients With Sacroiliac Joint Pain
Brief Title: Combined Corticosteroid Injections and Shockwave Therapy for Sacroiliac Joint Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Clinical Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B202405209
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Sacroiliac Joint Dysfunction; Sacroiliac Joint Pain
Keywords: Sacroiliac Joint Dysfunction; Sacroiliac joint pain; Steroid Injection; Extracorporeal shock wave therapy
MeSH Terms: interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Injection and shockwave Therapy (Experimental): Participants received ultrasound-guided sacroiliac joint corticosteroid injections (1 ml SHINCORT INJ 10 MG/ML + 1 ml 2% Xylocaine). One week later, they began a three-week course of weekly extracorporeal shockwave therapy sessions (intensity: low to moderate, adjusted based on patient tolerance; frequency: 5 Hz; 2000 shocks per session).
  Interventions: Drug: Corticosteroids Triamcinolone Acetonide; Device: extracorporeal shockwave
- Corticosteroid Injection and sham shockwave Therapy (Sham Comparator): Participants received ultrasound-guided sacroiliac joint corticosteroid injections (1 ml SHINCORT INJ 10 MG/ML + 1 ml 2% Xylocaine). One week later, they began a three-week course of weekly extracorporeal shockwave therapy sessions (intensity: minimum setting on the device; frequency: 5 Hz; 2000 shocks per session).
  Interventions: Drug: Corticosteroids Triamcinolone Acetonide; Device: extracorporeal shockwave(minimum intensity)

INTERVENTIONS:
Drug: Corticosteroids Triamcinolone Acetonide — ultrasound-guided sacroiliac joint corticosteroid injections (1 ml SHINCORT INJ 10 MG/ML + 1 ml 2% Xylocaine)
Device: extracorporeal shockwave — a three-week course of weekly extracorporeal shockwave therapy sessions (intensity: low to moderate, adjusted based on patient tolerance; frequency: 5 Hz; 2000 shocks per session)
  Arms: Corticosteroid Injection and shockwave Therapy
Device: extracorporeal shockwave(minimum intensity) — a three-week course of weekly extracorporeal shockwave therapy sessions (intensity: minimum setting on the device; frequency: 5 Hz; 2000 shocks per session)
  Arms: Corticosteroid Injection and sham shockwave Therapy

SUMMARY:
This study aims to investigate the combined use of corticosteroid injections and ESWT for SIJ pain.

DETAILED DESCRIPTION:
The most common primary cause of pain and stiffness from the SIJ is sacroiliac joint dysfunction. Currently, conservative treatments for SIJ dysfunction-related pain include oral anti-inflammatory pain medications, exercise therapy, physical therapy, and local injection therapies such as corticosteroids, dextrose, and platelet-rich plasma. Although there are multiple non-surgical options available for SIJ pain management, clear treatment guidelines have not yet been established. Among these options, intra-articular corticosteroid injections in the SIJ are frequently used by rehabilitation specialists in clinical practice, and their effectiveness in relieving pain from SIJ dysfunction has been demonstrated. However, the effects of corticosteroids in treating musculoskeletal-related diseases are typically short-term. Extracorporeal shock wave therapy (ESWT) has become increasingly common in the management of musculoskeletal conditions such as calcific tendinitis, tennis elbow, and plantar fasciitis, showing long-lasting benefits and inducing tissue repair responses that studies suggest may last up to two years. However, literature on ESWT for lower back pain is limited, and research on its use for SIJ pain is even rarer. Therefore, this study aims to investigate the combined use of corticosteroid injections and ESWT for SIJ pain, aiming to achieve rapid, short-term pain relief through corticosteroid injections, followed by potential long-term effects through ESWT.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain lasting for 3 months or more
* Pain VAS score of 4 or higher
* Three or more positive results in sacroiliac joint provocation tests
* At least 50% pain relief following ultrasound-guided sacroiliac joint injection with local anesthetic

Exclusion Criteria:

* Currently undergoing extracorporeal shockwave therapy in other areas
* Suspected pain caused by other lumbar spine or hip joint conditions (e.g., lumbar spine or disc disorders, radicular pain, spondylolisthesis/disc degeneration, hip arthritis)
* Presence of complex comorbidities, including trauma, systemic infections (e.g., fever, chills, night sweats), local sacroiliac joint infections, autoimmune diseases, or immunosuppression
* Sacroiliac joint injection therapy received within the past 6 months
* Contraindications for extracorporeal shockwave therapy (e.g., cancer or current/prior infections at the treatment site, pacemakers, pregnancy, epilepsy, or coagulation disorders caused by disease or medication)
* Impaired renal function preventing the administration of contrast agents for sacroiliac joint bone scanning

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
pain Visual Analogue Scale(VAS) | baseline, one week after treatment, and at 1, 3, and 6 months post-treatment
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. "0" means painless and "10" means extremely painful.

SECONDARY OUTCOMES:
Oswestry Disability Index, ODI | baseline, one week after treatment, and at 1, 3, and 6 months post-treatment
  The Oswestry Disability Index (ODI) was used to assess the degree of functional impairment caused by low back pain. The index consists of 10 items, each with 6 options scored from 0 to 5, representing varying levels of disability. A score of 0 indicates no disability, while a score of 5 indicates severe disability. The scores for all items are summed to obtain a total score, with a maximum possible score of 50, which is then expressed as a percentage.
Quantitative scintigraphy of the sacroiliac joints | baseline, 3 months post-treatment
  Quantitative scintigraphy of the sacroiliac joints is an imaging technique used to evaluate the sacroiliac joint, commonly employed to diagnose joint issues such as inflammation, joint lesions, or other pathological conditions causing pain. During the scanning process, a radiolabeled substance is typically injected into the body, which accumulates in areas of high bone activity, particularly those with inflammation or injury. This highlights metabolic activity or structural changes within the joint.

CONTACTS AND LOCATIONS:
Overall Officials: Liang cheng Chen, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General